CLINICAL TRIAL: NCT03608592
Title: Human Umbilical Cord Derived Mesenchymal Stem Cells Therapy in Acute Respiratory Distress Syndrome
Brief Title: Human Umbilical Cord Mesenchymal Stem Cells (MSCs) Therapy in ARDS
Acronym: ARDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lv Haijin, attending physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QHJH201804
Record Dates: First submitted 2018-07-10; First posted 2018-08-01 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: refractory acuter respiratory distress syndrome; mesenchymal stem cells; salvage therapy
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Suspensions; Saline Solution

STUDY DESIGN:
Intervention Model Description: A package of 100ml normal saline with 10^6/kg umbilical cord derived MSCs suspension will infused from central venous catheter.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UCMSCs group (Experimental): Intravenous infusion of 1million UCMSCs per kilogram body weight suspended in 100ml normal saline, infusion duration 30-60min.
  Interventions: Biological: umbilical cord derived mesenchymal stem cells (UCMSCs) suspension; Biological: normal saline

INTERVENTIONS:
Biological: umbilical cord derived mesenchymal stem cells (UCMSCs) suspension — Clinical grade human umbilical cord derived mesenchymal stem cells (passage 3-5) suspension are provided by biotherapy center of the third affiliated hospital of Sun Yat Sen University. Cells are made of suspension packages (60million cells in 100ml normal saline per bag) and infused intravenously in 2 hours.
Biological: normal saline — A bag of 100ml clinical grade normal saline are also provided by biotherapy center of the third affiliated hospital of Sun Yat Sen University.

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a devastating inflammatory and destructive disease in critical ill patients. Preclinical studies have shown a promising perspective of mesenchymal stem cells (MSCs) therapies in ARDS. But the safety and efficacy of umbilical cord MSCs (UCMSCs) have not yet been convinced in clinical trails. This study will explore the safety and life-rescue potential of UCMSCs in refracotry ARDS.

DETAILED DESCRIPTION:
This is a single arm study. According Berlin definition (2012), moderate or severe adult ARDS patients who fail to improve oxygenation (PaO2/FiO2 increase over 20%) in the first 24h or 8h after diagnosis will be enrolled. A salvage package of 10^6/kg suspended UCMSCs in 100ml normal saline or only 100ml normal saline will be infused through central venous catheter. Infusion associated events (IAEs) in 24 hours will be closely monitored. Compared with propensity score matched controls, mortality in 28 days as the primary outcomes. oxygenation index, ventilator parameters, lung injury biomarkers and clinical outcomes as secondary outcomes will be analyzed.

This is a revised trail from its previous registered pilot RCT, approved by Ethic Committe of Stem Cells Trails (ECSCT) of 3rd affiliated hospital of Sun Yat-Sen university

ELIGIBILITY:
Inclusion Criteria:

1. Aged≥18 years old;
2. Including all the criteria:

(1) Invasive ventilation, OI（PaO2/FiO2）<200; (2) PEEP≥8cmH2O; (3) Bilateral infiltration of lung in X-ray or CT; (4) In 1 week after onset; (5) Still OI<200 after protective ventilation or conservative fluid management.

Exclusion Criteria:

1. Any malignant disease;
2. Cardiogenic pulmonary edema;
3. Over 50% atelectasis either lung lobe in X-ray;
4. Pregnancy or perinatal or lactation;
5. Previous end stage respiratory disease;
6. More than 3 organs failure;
7. Liver failure with MELD(Model For End-Stage Liver Disease) score>40;
8. Stage III or IV pulmonary hypertension;
9. None invasive arterial and central venous catheter;
10. Concurrent deep venous thrombus or pulmonary embolism in 3 months;
11. Cerebral hernia;
12. More than 96 hours after ARDS onset.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Infusion associated events | From infusion beginning to the second day, 24 hours
  Incidence of prescribed adverse events or unprescribed events agreed by investigators and consultant .
Mortality | In 60 days after enrolled
  All cause mortality. Cause of death, exact survival status (death/survival) and time (days) will also be recorded

SECONDARY OUTCOMES:
Ventilation free days(VFDs) | From the day of UCMSCs use(day 0) to day 28
  The days without invasive ventilator support(at least 2 consecutive calendar days) in 28 days.
  If the ventilator weaned multiple times, VFDs is the sum of the days without ventilator support.
  If any of following occurring in 28 days, VFDs equals 0:
  1. The patient dies in 28 days;
  2. Ventilator never be weaned;
  3. Censored case with ventilator never being weaned.
Oxygenation index(OI) changes | From day 0 to day 7, each day
  The oxygenation index(OI)=partial pressure of oxygen in arterial blood(PaO2) divide inspiration fraction of oxygen(FiO2). OI is measured at day0, day1,day3,day7.
Lung injury score(LIS) | From day 0 to day 7, day0,1,3,7
  Murray lung injury scores (LIS) consist of the following 4 parts:
  A.Hypoxemia (PaO2/FiO2≥300, 225-299,175-224,100-174,<100, assigned 0,1,2,3,4 scores respectively); B.PEEP (cmH2O) (≤5,6-8,9-11,11-14,≥15, assigned 0,1,2,3,4 scores respectively) ; C.Compliance (ml/cmH2O)(≥80,60-79,40-59,20-39,≤19, assigned 0,1,2,3,4 scores respectively); D.Quadrants infiltrated in Chest X-Ray(CXR) (0,1,2,3,4, assigned 0,1,2,3,4 scores respectively).
  The total LIS score is obtained by dividing the total sum of points by the number of criteria present. For example, if only 3 criteria are answered to, the total sum is divided by 3 to reveal the final score.
  The LIS score ranges between 0 and 4, with scores closer to 4 indicating severe acute lung injury.
Positive end expiratory pressure(PEEP) | From day 0 to day 7, each day
  Monitored by ventilator and recorded per hour, obtain the average value of the day. unit-cmH20
Plateau pressure(Pplat) | From day 0 to day 7, each day
  Monitored by ventilator in one inspiration pause, measured 4 times a day. Record the average value of the day. unit-cmH20
Driving pressure | From day 0 to day 7, each day
  Calculate the driving pressure by Pplat minus PEEP, measured 4 times a day. Record the average value of the day. unit-cmH20
Static compliance | From day 0 to day 7, each day
  Calculate the static compliance by the following formula:
  static compliance=tidal volume/(Pplat-PEEP), unit-ml/cmH2O

OTHER OUTCOMES:
Epithelial injury biomarker-KL6 | From day 0 to day 7, day0, 1,3,7
  Detect Krebs von den Lungen-6(KL6) level in bronchoalveolar fluid (BALF), unit-U/ml
Endothelial injury biomarker-Ang2 | From day 0 to day 7, day0, 1,3,7
  Detect the angiopoietin (Ang2) level in plasma, unit-pg/ml
Tumor necrosis factor a(TNFa) | From day 0 to day 7, day0, 1,3,7
  Detect the TNFa in plasma and in BALF, unit-pg/ml
Interleukin 8(IL8) | From day 0 to day 7, day0, 1,3,7
  Detect the IL8 in plasma and in BALF, unit-pg/ml
Interleukin 6(IL6) | From day 0 to day 7, day0, 1,3,7
  Detect the IL6 in plasma and in BALF, unit-pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Huimin Yi, Principal Investigator — The 3rd affiliated hospital of Sun Yat-sen University
Locations (1):
- Huimin Yi, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided